CLINICAL TRIAL: NCT01335867
Title: A Phase II, Double-Blind, Placebo-Controlled, Pilot Trial of Vigabatrin for the Treatment of Cocaine and Alcohol Dependence
Brief Title: Vigabatrin for Cocaine and Alcohol Dependence
Acronym: VGB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: interim analysis of efficacy completed and termination recommended
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812864; P50DA012756 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Alcoholism; Cocaine Dependence
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders | interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vigabatrin (Experimental): Vigabatrin titrated to 3 grams daily for 8 weeks
  Interventions: Drug: Vigabatrin
- Placebo (Placebo Comparator): Identical placebo daily for three weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vigabatrin — Vigabatrin escalated to 3 grams daily for 8 weeks
  Other Names: Sabril
  Arms: Vigabatrin
Drug: Placebo — Placebo pills
  Other Names: placebo vigabatrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of vigabatrin at reducing drug and alcohol use in individuals addicted to cocaine and alcohol. Vigabatrin is approved for the treatment of seizures. It has not been proven to be effective for the treatment of alcohol or cocaine dependence.

DETAILED DESCRIPTION:
The hypotheses in the proposed study will be tested with a 2-group design to assess the efficacy of vigabatrin compared to placebo. We will follow NIAAA's COMBINE Medical Management (MM) manual in weekly dispensing medications, safety checks and medication adherence. The psychosocial treatment will be Cognitive Behavioral Coping Skills Therapy (CBT). Subjects will be 60 men and women with current DSM-IV diagnoses of both cocaine and alcohol dependence who will be randomized to vigabatrin or placebo (30 subjects per group). All subjects will receive weekly sessions of CBT. The study length for each subject is comprised of a1-3 weeks of screening and baseline evaluations, an 8-week double-blind, placebo-controlled trial with CBT (medication phase), and one follow-up visit 12 weeks after starting study medication.

Study medication will be initiated in Week 2. The research physician will explain the dosing regimen and subjects will be randomly assigned to receive either vigabatrin or identical placebo tablets. Subjects will receive 1 gram of vigabatrin or identical placebo tablets on medication days 1-3 then 1.5 grams or identical placebo tablets on days 4-7. The dose ids increased to 2 grams in week 2, 3 grams in weeks 4-7 and then reduced to 2 grams days 50-53, and to 1 gram on days 54-56

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, 18 years of age or older.
2. Meets DSM-IV criteria for current diagnoses of cocaine and alcohol dependence, determined by the SCID-IV.
3. Used cocaine in the past 30 days and used no less than $200 of cocaine in a consecutive 30 day period over the 90 day period prior to intake. Meets the following drinking criteria as measured by the Timeline Followback (TLFB) (Sobell 1995) a drank within 30 days of intake day, b. reports a minimum of 48 standard alcoholic (avg. 12 drinks/wk) in a consecutive 30-day period over the 90-day period prior to starting intake (i.e., a minimum of 40% days drinking), and c. has 2 or more days of heavy drinking (defined as greater than 4 drinks per day in males and greater than 3 drinks per day in females) in this same pre-treatment period.
4. Three consecutive days of abstinence from alcohol directly prior to the day of randomization, determined by self-reports and confirmed by negative breathalyzer tests, and a Clinical Institute Withdrawal Scale for Alcohol (CIWA-AR) (Sullivan and Sellers 1989) score below eight. Subjects will be given 2 additional weeks beyond the screening week to attain the appropriate period of alcohol abstinence prior to randomization.
5. Have a verifiable address of principal residence, lives a commutable distance from the TRC and agrees to attend all research visits including follow-up visits.
6. Speaks, understands, and prints in English
7. Ability to give informed consent

Exclusion Criteria:

1. Meets DSM IV criteria for dependence on any substance other than cocaine and alcohol (except nicotine and cannabis), determined by the SCID. Needs treatment with any psychoactive medications including any anti-seizure medications (with the exception of diphenhydramine used sparingly, if necessary, for sleep).
2. Meets current or lifetime DSM-IV criteria for schizophrenia or any psychotic disorder or organic mental disorder. Subject meets current DSM-IV diagnosis of any other clinically significant psychiatric disorder that will interfere with study participation as determined by the principal investigator.
3. Has evidence of a history of significant hematological, pulmonary, endocrine, cardiovascular, renal or gastrointestinal disease.
4. Severe physical or medical illnesses such as AIDS, active hepatitis, significant hepatocellular injury as evidenced by elevated total bilirubin levels (>1.3 mg/dl), or elevated levels (over 4.5x normal) of aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT). Patients with Gilberts Syndrome will not be excluded.
5. Use of an investigational medication in the 30 days prior to randomization.
6. History of prior treatment with vigabatrin
7. History of prior treatment with drugs with known retinotoxicity
8. History of visual field defects or predisposing factors, including glaucoma, severe myopia, retinal disorders, cataracts, diabetes, or uncontrolled hypertension.
9. Is female and tests positive on a pregnancy test, is contemplating pregnancy in the next 6 months, is nursing, or is not using an effective contraceptive method (if relevant). Acceptable methods of contraception include barrier methods (diaphragm or condom with spermicide, female condom), intrauterine progesterone contraceptive system, levonorgrestrel implant, and medroxyprogesterone acetate contraceptive injection, copper IUD, vaginal contraceptive film, cervical cap, contraceptive foam, hormonal vaginal contraceptive ring (NuvaRing®) or oral contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Kampman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: University of Pennsylvania Center for Studies of Addictions — http://www.med.upenn.edu/csa/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vigabatrin | Placebo
Started | 16 | 16
Completed | 9 | 12
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vigabatrin | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (7.97) | 48 (6.81) | 47 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Cocaine Use
Description: The primary outcome measure for reduction in cocaine use will be the number of benzoylecgonine (BE) negative urine samples. The main outcome is the number of participants in each group who reported all BE negative urine samples in the last three weeks of the trial.
Time Frame: last 3 weeks of the trial
Measure: Number; unit: participants
Groups:
- Vigabatrin: Vigabatrin: Vigabatrin escalated to 3 grams daily for 12 weeks
Arm/Group | Vigabatrin | Placebo
Number analyzed (Participants) | 16 | 16
participants | 0 | 2
Statistical Analysis 1: Comparison: Vigabatrin vs Placebo; Test type: Superiority; p = .14, Chi-squared

2. Primary Outcome: Proportion of Heavy Drinking Days
Description: The primary outcome measure for reduction in alcohol use will be recorded using the Timeline Followback method.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: proportion of heavy drinking days
Arm/Group | Vigabatrin | Placebo
Number analyzed (Participants) | 16 | 16
proportion of heavy drinking days | .26 (.18) | .20 (.25)

3. Secondary Outcome: Measures of Cocaine Craving
Description: Measures of cocaine craving at the end of the trial will be measured using the Brief Substance Craving Ccale. Craving intensity + Craving frequency + Craving Duration each measured on a 4 point scale. Sum of the three scales was overall craving composite. Higher numbers meaning greater craving. Maximum score 12 minimum 0.
Time Frame: 8 weeks
Population: subjects receiving vigabatrin or placebo who were available at the end of the trial to provide data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Vigabatrin: vigabatrin 3 grams daily for 12 weeks
- Placebo: placebo capsules
Arm/Group | Vigabatrin | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 1.44 (2.3) | 0.38 (1.1)
Statistical Analysis 1: Comparison: Vigabatrin vs Placebo; Test type: Superiority; p = .24, t-test, 2 sided

4. Secondary Outcome: Disease Severity and Improvement
Description: Number of subjects in each group rated as improved or very much improved at the end of the trial
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Vigabatrin: Vigabatrin titrated to 3 grams daily for 12 weeks
  Vigabatrin: Vigabatrin escalated to 3 grams daily for 8 weeks
- Placebo: Identical placebo daily for 12 weeks
  Placebo: Placebo pills
Arm/Group | Vigabatrin | Placebo
Number analyzed (Participants) | 16 | 16
Participants | 5 | 2
Statistical Analysis 1: Comparison: Vigabatrin vs Placebo; Test type: Superiority; p = .20, Chi-squared

5. Secondary Outcome: Cocaine Withdrawal Severity
Description: Measure of cocaine withdrawal severity will include Cocaine Selective Severity Assessment scores. Minimum score is 0 Maximum score is 119 Higher score is indicative of worse cocaine withdrawal symptoms.
Time Frame: 8 weeks
Population: subjects receiving vigabatrin or placebo who were available at the end of the trial to provide data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vigabatrin | Placebo
Number analyzed (Participants) | 10 | 11
score on a scale | 8.0 (8.1) | 6.5 (6.8)
Statistical Analysis 1: Comparison: Vigabatrin vs Placebo; Test type: Superiority; p = .64, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Vigabatrin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 10/16 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vigabatrin (N=16) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 2 | 0
Headache (General disorders) | 2 | 0
Dry Mouth (General disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
URI Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal Congestion (Skin and subcutaneous tissue disorders) | 0 | 2
Sore Knees (Musculoskeletal and connective tissue disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No